CLINICAL TRIAL: NCT03495245
Title: Development of a Serum Biomarker-Based Approach to Monitor Opioid Adherence and Minimize Substance Misuse in Chronic Pain Management
Brief Title: Identification of Potential Biomarkers for Pain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rowan University (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Venkat Venkataraman, PhD, Assistant Professor, Rowan University
Other Study IDs: Pro2017001740
Record Dates: First submitted 2018-01-18; First posted 2018-04-11 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Fibromyalgia
Keywords: pain; opioid; fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood will be collected from the subjects. Serum and plasma will be obtained from the samples and retained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opioid Usage: Patients that are currently diagnosed with fibromyalgia and taking opioids.
- No Opioid Usage: Patients that are currently diagnosed with fibromyalgia and are not taking opioids.

SUMMARY:
The study investigates the potential of using serum biomarkers to assess pain in fibromyalgia patients.

DETAILED DESCRIPTION:
At the heart of the opioid epidemic is the lack of an objective measure of pain, which will help evaluate the validity of the patients' perception that the current dosage of opioid is sufficient of insufficient to alleviate pain. This study will test the quantifiable proteins such as S100B and BDNF will serve as objective measures (biomarkers) of pain.

Fibromyalgia patients will be recruited into two groups-- one that uses opioids and the other that does not. Blood will be collected every 6 months for two years. The serum will be used to assay for levels of S100B and BDNF, The pressure-pain threshold (PPT) data, as part of standard of care, will also be collected. Correlation will the be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Fibromyalgia

Exclusion Criteria:

* Evidence of a history of substance abuse, neurological or oncologic disease, ischemic heart disease, kidney or hepatic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are seen at the NeuroMusculoskeletal Institute at Rowan University School of Osteopathic Medicine.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum protein levels as a marker for pain | 2-4 years
  Serum proteins will be assayed from patients. The correlation between the serum levels and the visual analog pain scale will be determined.
  0 on the visual analog pain scale represents that their is no pain. 10 on the visual analog pain scale represents severe pain.

SECONDARY OUTCOMES:
Determine if correlation may be established between impact of fibromyalgia and opioid doses | 2-4 years
  The prescribed opioid doses, if effective, will be expected to reduce/maintain the scores from the Revised Fibromyalgia Impact Questionnaire. Correlations will be determined through established statistical methods.
  The results from the FIQR can estimate the fibromyalgia severity and impact.
Determine if correlation may be established between sleep index and opioid doses | 2-4 years
  The prescribed opioid doses, if effective, will be expected to reduce/maintain the scores from the Sleep Questionnaire. Correlations will be determined through established statistical methods.
  This questionnaire can help determine the overall quality of person's sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Venkateswar Venkataraman, PhD, Principal Investigator — Rowan University School of Osteopathic Medicine
Locations (1):
- Rowan University School of Osteopathic Medicine, Stratford, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.